CLINICAL TRIAL: NCT05145101
Title: Immunogenicity of the Currently Recommended Pneumococcal Vaccination Schedule in Patients With Chronic Lymphocytic Leukaemia.
Brief Title: Pneumococcal Vaccination in Patients With Chronic Lymphocytic Leukaemia
Acronym: Pneumo-CLL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannah Garcia Garrido (Other)
Responsible Party: Sponsor-Investigator, Hannah Garcia Garrido, Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: W20_197#20.228
Record Dates: First submitted 2021-11-18; First posted 2021-12-06 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Pneumococcal Infections; Chronic Lymphocytic Leukemia; Vaccine-Preventable Diseases; Invasive Pneumococcal Disease, Recurrent Isolated
MeSH Terms: conditions — Pneumococcal Infections; Leukemia, Lymphocytic, Chronic, B-Cell; Vaccine-Preventable Diseases; IRAK4 Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes

INTERVENTIONS:
Biological: Prevnar13 — Patients receive one dose of Prevenar13 followed by one dose of Pneumovax23 2 months later
  Other Names: Pneumovax23

SUMMARY:
In this study the antibody response after vaccination with the 13-valent pneumococcal conjugated vaccine (PCV13) followed 2 months later by the 23-valent polysaccharide vaccine (PPSV23) in adults with chronic lymphocytic leukemia will be investigated.

DETAILED DESCRIPTION:
Background Patients with chronic lymphocytic leukaemia (CLL) are at increased risk of both invasive pneumococcal disease (IPD) and community acquired pneumonia (CAP) caused by Streptococcus pneumoniae. Therefore, international guidelines recommend pneumococcal vaccination for all CLL patients, preferably before initiation of treatment. The recommended vaccination schedule consists of Prevenar13®, a 13-valent pneumococcal conjugated vaccine (PCV13) followed 2 months later by Pneumovax23, a 23-valent polysaccharide vaccine (PPSV23).

The immunological efficacy of this sequential vaccination schedule in CLL patients is unknown. Previous studies have only investigated responses to either PCV13 or PPSV23 alone. Responses to PPSV23 alone are poor in CLL patients. Responses to the 7-valent pneumococcal conjugated vaccine (PCV7) or PCV13 are higher compared to responses to PPSV23, but lower compared to responses in healthy individuals. More advanced disease stage and lower baseline IgG negatively influence responses to vaccination.

The aim of this observational cohort study is to assess the immunogenicity of the currently recommended vaccination schedule of PCV13 followed by PPSV23 in CLL patients.

2. Methods Study design and population As part of routine care, all adult CLL patients naïve to pneumococcal vaccination and cared for in the Amsterdam UMC-location AMC, Flevoziekenhuis, HagaZiekenhuis, Elisabeth-TweeSteden Hospital, Noordwest Ziekenhuisgroep, Albert Schweitzer Hospital and Ikazia Hospital receive one dose of Prevenar13® followed by one dose of Pneumovax23® 2 months later. According to the current local standard of care for immunosuppressed individuals, the response to vaccination will be assessed by measuring pneumococcal antibody levels before and 4-8 weeks after vaccination.

After obtaining informed consent clinical data will be collected by a trained medical student, nurse or research assistant according to a standardized electronic case report form (Castor EDC). Variables included in the case report form are: age, sex, smoking behaviour, Rai stage (I/II/III), past or ongoing chemotherapy, ongoing steroid treatment, past or ongoing therapy with a monoclonal anti-CD20 antibody (and date of last infusion), baseline total IgG level, baseline lymphocyte count, baseline haemoglobin level, baseline platelet level, baseline pneumococcal IgG levels, post-vaccination pneumococcal IgG levels, date of PCV and PPSV23 vaccine administration, date of antibody measurements, comorbidities (Charlson comorbitiy index).

Laboratory methods and definitions Serotype-specific pneumococcal immunoglobulin G (IgG) concentrations to 5 pneumococcal serotypes shared across both vaccines (6B, 9V, 14, 19F, 23F) and 4 serotypes unique to PPSV23 (8, 15B, 20, 33F) will be determined in the immunology laboratory of the UMC Utrecht. A validated multiplex immunoassay will be used (Luminex® technology). Serologic response will be defined as a ≥4-fold increase in serotype specific anti-pneumococcal IgG for ≥70% of measured. Serologic protection will be defined as an antibody concentration ≥1.3 mcg/ml for ≥70% of all measured serotypes, according to the definition of the American Academy of Allergy, Asthma & Immunology. In addition, because most previous studies used the WHO cut-off for protection in infants (≥0.35mcg/ml) data will also be analyzed by the infant correlate of protection to be able to compare the results with previous studies.

ELIGIBILITY:
Inclusion Criteria:

* CLL
* Age >17
* Naive to pneumococcal vaccination

Exclusion Criteria:

* Not able/willing to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: As part of routine care, all adult CLL patients naïve to pneumococcal vaccination must receive one dose of Prevenar13® followed by one dose of Pneumovax23® 2 months later. According to the current local standard of care for immunosuppressed individuals, the response to vaccination will be assessed by measuring pneumococcal antibody levels before and 4-8 weeks after vaccination
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-05-07 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
serologic response rate | 1-2 months after vaccination schedule
  Proportion of participants with a ≥4-fold increase in serotype specific anti-pneumococcal IgG for ≥6/9 serotypes

SECONDARY OUTCOMES:
Serologic protection rate | 1-2 months after vaccination
  Antibody concentration ≥1.3 mcg/ml for ≥6/9 serotypes
Geometric mean concentrations of serotype specific anti-pneumococcal IgG for 9 pneumococcal serotypes | Month 0, month 4

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC Locatie AMC, Amsterdam-Zuidoost, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT05145101/Prot_SAP_000.pdf